CLINICAL TRIAL: NCT05169489
Title: A Phase 1/2 Study of bbT369, a Dual Targeting CAR T Cell Drug Product With a Gene Edit, in Relapsed and/or Refractory B Cell Non-Hodgkin's Lymphoma (NHL)
Brief Title: A Study of bbT369 in Relapsed and/or Refractory B Cell Non-Hodgkin's Lymphoma (NHL)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC-403
Record Dates: First submitted 2021-12-11; First posted 2021-12-27 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
Keywords: CAR T; CART; CAR-T; Cell therapy; Lymphoma; Diffuse large B cell lymphoma (DLBCL); Primary mediastinal (thymic) large B cell lymphoma (PMBCL); High-grade B cell lymphoma (HGBCL); Follicular lymphoma (FL) 3b; DLBCL transformed from FL; NHL; Non hodgkin's; Dual targeting; Gene edit; T cell; CD20; CD79a; CBLB; Non-hodgkin's; Non-hodgkin
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- bbT369 Experimental Arm (Experimental): Open label, single arm treatment with bbT369
  Interventions: Biological: bbT369

INTERVENTIONS:
Biological: bbT369 — bbT369 is a genetically modified autologous T cell immunotherapy product consisting of T cells that are transduced with a single lentiviral vector (LVV) to express anti-CD79a and anti-CD20 chimeric antigen receptors (CARs) and transfected with an mRNA encoding the CBLB-targeting megaTAL enzyme to edit the CBLB gene, suspended in a cryopreservative solution.

SUMMARY:
This non-randomized, open label, multi-site, first-in-human, Phase 1/2 study CRC-403 will evaluate the safety and efficacy of bbT369 in subjects with relapsed and/or refractory B cell non-Hodgkin's lymphoma (NHL).

A long-term follow-up (LTF-01 [NCT06798298]) is planned, in which subjects who received bbT369 will be followed for up to 15 years after drug product infusion to evaluate for safety and continued efficacy.

DETAILED DESCRIPTION:
Former Sponsor 2seventy bio

The trial was intended to be a Phase 1/2 trial, but no participants were enrolled in Phase 2, consequently the study was terminated in Phase 1.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age at the time of signing informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Diagnosis of B-cell NHL according to WHO 2017 classification or WHO 2016 classification where applicable:

  1. DLBCL (germinal center B cell [GCB] or activated B cell [ABC] type or not otherwise specified [NOS])
  2. HGBCL (with MYC and BCL2 and/or BCL6 rearrangements or NOS)
  3. PMBCL
  4. FL 3b
  5. DLBCL transformed from FL
* Participants must have relapsed or refractory (r/r) B cell NHL after autologous stem cell transplant (ASCT) or at least 2 prior lines of therapy including an anti-CD20 monoclonal antibody and an anthracycline containing chemotherapy regimen. Note: participants with DLBCL transformed from FL must have r/r disease after ASCT or at least 2 prior therapies following transformation irrespective of therapeutic agents.
* At least 1 FDG-avid lesion per Lugano Classification criteria at time of enrollment.

Exclusion Criteria:

* Treatment with any investigational cellular therapy prior to enrollment. Treatment with an approved anti-CD19 CAR T cell therapy in an investigational setting may be permitted after discussion with and approval of the Sponsor.
* Progression within 6 weeks of prior anti-CD19 CAR T cell therapy.
* Residual toxicities or end-organ damage to vital organs from prior therapy that could put a subject at undue risk based on Investigator's assessment. Toxicities related to prior cytokine release syndrome (CRS) or neurotoxicity must be resolved.
* If a subject has received prior anti-CD19 CAR T therapy, development of ≥ Grade 3 CAR T related CRS or ≥ Grade 3 neurotoxicity that in the opinion of the Investigator would cause unacceptable risk of toxicity to the subject upon treatment with bbT369.
* Primary central nervous system (CNS) lymphoma or a history or presence of clinically relevant CNS pathology.
* Active autoimmune disease requiring systemic immunosuppressive and/or cytotoxic therapy within the past two years.
* Treatment with any prior anti-CD79a therapy.
* Previous history of an allogeneic bone marrow transplantation. Autologous stem cell transplantation (ASCT) is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Phase 1: Incidence of safety events including: adverse events (AEs), adverse events of special interest (AESIs), and dose limiting toxicities (DLTs) | Day 1 through Month 24

SECONDARY OUTCOMES:
Phase 1: Rates of disease-specific response criteria including complete response rate(CRR), partial response rate(PRR), stable disease rate(SDR), and progressive disease rate(PDR) according to the Lugano 2014 response criteria as assessed by Investigator | Day 1 through Month 24
Phase 1: Overall Response Rate (ORR) according to the Lugano 2014 response criteria as assessed by Investigator | Day 1 through Month 24
Phase 1: Time to response (TTR) | Day 1 through Month 24
Phase 1: Time to complete response (TCR) | Day 1 through Month 24
Phase 1: Time to next treatment for B Cell NHL (TTNT) | Day 1 through Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (4):
- United States (4):
  - Stanford Cancer Institute, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Sarah Cannon, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes